CLINICAL TRIAL: NCT04213261
Title: A Pivotal Phase 3 Study of FCX-007 (Genetically-Modified Autologous Human Dermal Fibroblasts) for Recessive Dystrophic Epidermolysis Bullosa
Brief Title: A Study of FCX-007 for Recessive Dystrophic Epidermolysis Bullosa
Acronym: DEFI-RDEB
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FI-EB-002; R01-7289-01 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2019-12-02; First posted 2019-12-30 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: RDEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: Intra-patient Randomized, Controlled, Open-label, Multi-center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts (Experimental): Intra-subject randomized (paired wounds in each subject receive experimental treatment, FCX-007, or remain untreated). Up to three target wound pairs will be identified for each subject. Following pairing, target wounds will be randomly assigned as the treatment wound (FCX-007 is administered) or control wound. Subjects will receive intradermal injections of FCX-007 in each specified treatment wound in two or more treatment sessions. The first treatment session occurs at Day 1 and the second at Week 12/Month 3. Additional treatment sessions may occur at Week 24/Month 6 and Week 36/Month 9 when unclosed treatment wounds may be re-treated, and unclosed control wounds may be treated.
  Interventions: Biological: FCX-007 (dabocemagene autoficel; see below for FCX-007 description)

INTERVENTIONS:
Biological: FCX-007 (dabocemagene autoficel; see below for FCX-007 description) — FCX-007 is comprised of fibroblasts isolated from the subject's skin biopsies which are genetically corrected with the full length COL7A1 gene encoding for type VII collagen.

SUMMARY:
The purpose of this study is to determine whether administration of FCX-007 in addition to standard of care improves wound healing as compared to standard of care alone (control) in children, adolescents, and adults with Recessive Dystrophic Epidermolysis Bullosa.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
DEFI-RDEB is a multi-center, intra-patient randomized, controlled, open-label, Phase 3 study of FCX-007 for the treatment of persistent non-healing and recurrent RDEB wounds in approximately 24 subjects. Each subject will serve as his/her own control. Each subject's target wounds will be paired then randomized to receive FCX-007 (treatment wound) or remain untreated (control wound). Up to three target wound pairs will be identified for each subject.

Subjects will receive intradermal injections of FCX-007 in each specified treatment wound in two or more treatment sessions. The first treatment session occurs at Day 1 and the second at Week 12/Month 3. Additional treatment sessions may occur at Week 24/Month 6 and Week 36/Month 9 when unclosed treatment wounds may be re-treated, and unclosed control wounds may be treated. Safety and efficacy assessments will occur at scheduled intervals through Week 48/Month 12, when the treatment period is completed, and a long-term safety follow-up period (through 15 years) commences for subjects who have received one or more FCX-007 injections.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥2 years of age at the Screening visit.
* Clinical diagnosis of RDEB with confirmation of COL7A1 genetic mutation.

Key Exclusion Criteria:

* Medical instability limiting ability to travel to the investigative site.
* Active infection with human immunodeficiency virus, hepatitis B or hepatitis C.
* The presence of COL7 antibodies.
* Evidence of systemic infection.
* Evidence or history of squamous cell carcinoma at the site to be injected.
* Evidence of or history of metastatic squamous cell carcinoma.
* Known allergy to any of the constituents of the product.
* Female who is pregnant or breastfeeding.
* Receipt of a chemical or biological intervention for the specific treatment of RDEB in the past three (3) months prior to screening or anticipated/planned during the screening and treatment period for this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2037-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Dell Children's Medical Group, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: wound
Groups:
- FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts; Control (no Treatment): All subjects, intra-subject randomized (paired wounds in each subject receive experimental treatment, FCX-007, or remain untreated). Up to three target wound pairs will be identified for each subject. Following pairing, target wounds will be randomly assigned as the treatment wound (FCX-007 is administered) or control wound. Subjects will receive intradermal injections of FCX-007 in each specified treatment wound in two or more treatment sessions. The first treatment session occurs at Day 1 and the second at Week 12/Month 3. Additional treatment sessions may occur at Week 24/Month 6 and Week 36/Month 9 when unclosed treatment wounds may be re-treated, and unclosed control wounds may be treated.
  FCX-007 (dabocemagene autoficel): FCX-007 is comprised of fibroblasts isolated from the subject's skin biopsies which are genetically corrected with the full length COL7A1 gene encoding for type VII collagen.
Period: Overall Study
Arm/Group | FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts | Control (no Treatment)
Started | 6; 13 wound | 6; 13 wound
Completed | 6; 13 wound | 6; 13 wound
Not Completed | 0; 0 wound | 0; 0 wound

BASELINE CHARACTERISTICS:
Arm/Group | FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (16.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Wound Closure of the First Wound Pair at Week 24
Description: Complete wound closure of the first wound pair (treated vs. control)
Time Frame: Week 24
Measure: Number; unit: wound
Units Other Than Participants: wound
Groups:
- FCX-007 Treated Success: Primary wound treated with FCX-007 with complete wound closure at serial assessments at Week 22 and 24
- Control Success: Primary control wound with complete wound closure at serial assessments at Week 22 and 24
Arm/Group | FCX-007 Treated Success | Control Success
Number analyzed (Participants) | 6 | 6
Number analyzed (wound) | 6 | 6
wound | 1 | 0

2. Secondary Outcome: Complete Wound Closure of the First Wound Pair at Week 12
Description: Complete wound closure of first wound pair (treated vs. control)
Time Frame: Week 12
Measure: Number; unit: wound
Units Other Than Participants: wound
Groups:
- FCX-007 Treated Success: Primary wound treated with FCX-007 with complete wound closure at Week 12
- Control Success: Primary control wound with complete wound closure at Week 12
Arm/Group | FCX-007 Treated Success | Control Success
Number analyzed (Participants) | 6 | 6
Number analyzed (wound) | 6 | 6
wound | 1 | 1

3. Secondary Outcome: Complete Wound Closure of All Wound Pairs at Week 24
Description: Complete wound closure
Time Frame: Week 24
Measure: Number; unit: wound
Units Other Than Participants: Wounds
Groups:
- FCX-007 Treated Success: All treated with FCX-007 with complete wound closure at Week 24
- Control Success: Primary control wound with complete wound closure at Week 24
Arm/Group | FCX-007 Treated Success | Control Success
Number analyzed (Participants) | 6 | 6
Number analyzed (Wounds) | 13 | 13
wound | 1 | 2

4. Secondary Outcome: Complete Wound Closure of All Wound Pairs at Week 12
Description: Complete wound closure
Time Frame: Week 12
Measure: Number; unit: wound
Units Other Than Participants: wound
Groups:
- FCX-007 Treated Success: All treated with FCX-007 with complete wound closure at Week 12
Arm/Group | FCX-007 Treated Success | Control Success
Number analyzed (Participants) | 6 | 6
Number analyzed (wound) | 13 | 13
wound | 1 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs), regardless of relationship to FCX-007, are those reported from start of treatment to end of treatment period (Week 48)
Description: All treatment-emergent AEs, regardless of relationship to FCX-007, are reported. AEs at a treated wound were to be described and coded as injection site reactions, AEs at other wounds (including but not limited to control wounds) were described without specific reference to injection-site. Only a single interventional group is included, inclusive of all study participants who have received FCX-007 and had at least one control wound.
Arm/Group | FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts (N=6)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCX-007 COL7A1 Genetically-Corrected Autologous Fibroblasts (N=6)
Tachycardia (Cardiac disorders) | 1 (1)
Injection site pain (General disorders) | 1 (2)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT04213261/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT04213261/SAP_003.pdf